CLINICAL TRIAL: NCT00281866
Title: Genotypic-Based Pharmacodynamic Evaluation of Erlotinib (Erlotinib (Tarceva™, OSI Pharmaceuticals, Uniondale, NY) in Patients With Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Erlotinib in Treating Patients With Metastatic and/or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: J0520 CDR0000452784; R21CA109283 (NIH); P30CA006973 (NIH); JHOC-J0520; JHOC-05042801
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with recurrent and/or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the relationship between response rate and number of CA repeats in intron 1 of the epidermal growth factor receptor (EGFR) in patients with metastatic and/or locally recurrent squamous cell carcinoma of the head and neck (SCCHN) treated with the EGFR inhibitor erlotinib hydrochloride.

Secondary

* Determine the relationship between the number of CA repeats in intron 1 of the EGFR gene and time to disease progression and survival in patients treated with this drug.
* Determine cutaneous and other toxicities of erlotinib hydrochloride in patients with different numbers of CA repeats in intron 1 of the EGFR gene.
* Compare the degree of p27 upregulation and EGFR phosphorylation in skin biopsy samples in patients with different numbers of CA repeats in intron 1 of the EGFR genes treated with this drug.
* Determine the relationship between erlotinib hydrochloride exposure (utilizing total and unbound erlotinib hydrochloride concentrations) and outcome, toxicity, and pharmacodynamic effects (upregulation of p27) in patients with different numbers of CA repeats.

OUTLINE: This is a multicenter study. Patients are stratified according to genotype of intron 1 of the epidermal growth factor receptor (16/16 vs 16/20 or 20/20).

Patients receive oral erlotinib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Metastatic and/or locally recurrent disease
  * No undifferentiated and nonkeratinizing carcinomas, including lymphoepitheliomas of all locations, as well as tumors of the parotid gland

    * WHO Type I squamous cell carcinoma of the nasopharynx are allowed
* Incurable with surgery or radiotherapy
* Measurable disease, defined as ≥ 1 target lesion ≥ 20 mm OR ≥ 10 mm on spiral CT scan

  * If the only site of measurable disease is in a previously irradiated area, the patient must have documented progressive disease by tomography or biopsy-proven residual carcinoma
* No symptomatic brain metastases that are not stable, are not adequately controlled with fixed-dose oral steroids, are potentially life-threatening, or have required radiotherapy within the last 14 days

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Predicted life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and/or ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must practice effective contraceptive measures
* No other prior malignancy within the past 3 years except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* No active or uncontrolled infection or other serious illnesses or medical conditions
* No history of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than two prior chemotherapy regimens for locally recurrent and/or metastatic disease
* Prior induction chemotherapy or chemoradiotherapy with curative intent for local disease allowed provided patient has received no more than two prior chemotherapy regimens for recurrent disease
* Prior therapy must have been completed a minimum of 14 days prior to study AND patient has recovered
* No prior molecular-directed therapies, such as tyrosine kinase inhibitors and/or monoclonal antibodies
* At least 14 days must have elapsed between the end of radiotherapy and study registration and recovered
* At least 14 days since prior surgery AND wound healing has occurred
* At least 7 days since prior herbal extracts and tinctures with CYP3A inhibitory activity, including any of the following:

  * Hydrastis canadensis (goldenseal)
  * Uncaria tomentosa (cat's claw)
  * Echinacea angustifolia roots
  * Trifolium pratense (wild cherry)
  * Matricaria chamomilla (chamomile)
  * Glycyrrhiza glabra (licorice)
  * Dillapiol
  * Naringenin
* No other concurrent anticancer therapy or other investigational agents
* No concurrent administration of any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampicin
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
  * CYP3A inhibitors (e.g., itraconazole)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Relationship between response rate and number of CA repeats in intron 1 of the EGFR

SECONDARY OUTCOMES:
Time to disease progression
Survival
Toxicity
Compare the degree of p27 upregulation and EGFR phosphorylation in skin biopsy samples
Relationship between erlotinib hydrochloride exposure and outcome, toxicity, and pharmacodynamic effects

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Gibson, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States
- Hospital Universitario 12 de Octubre, Madrid, Spain